CLINICAL TRIAL: NCT01506583
Title: Clinical Evaluation of QFlu Combo Test
Acronym: QFlu
Status: Completed | Type: Observational
Sponsor: Cellex, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Cellex002; 2R44AI082728-02 (NIH)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Cough; Myalgia; Nasal Obstruction; Sore Throat; Headache; Fatigue; Fever
Keywords: cough; myalgia; nasal obstruction; sore throat; headache; fatigue; feverishness; Patients who exhibit flu-like symptoms during a flu season, including cough, myalgia, nasal obstruction, sore throat, headache, fatigue, and/or feverishness.
MeSH Terms: conditions — Cough; Myalgia; Nasal Obstruction; Pharyngitis; Headache; Fatigue; Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples were retained in case that the testing needs to be repeated. They are to be discarded 12 months after the study is completed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- General population: This group of participants is primarily an out-patient population.
- In-patient population: This group of participants is primarily an in-patient population.
- Pediatric Group: Participants in this group are children 18 years or younger.

SUMMARY:
Currently effective antivials for influenza treatment are two influenza viral neuraminidase inhibitors, oseltamivir (Tamiflu) and zanamivir (Relenza). Resistance to these drugs is reflected by reduced susceptibility of viral neuraminidase to these drugs. The hypothesis is that the signal ratio of two reagents (with or without a single concentration of the drug) correlates the IC50 value, an accurate measurement of drug resistance but impractical for clinical use.

DETAILED DESCRIPTION:
The study design is to collect samples from participants. A portion of the sample is used for drug resistance detection using the test (QFlu Combo Test) under investigation. The remaining portion of the sample is used for culture. The culture positive samples are used for determination of IC50 values, which is used as a gold standard for defining whether a virus isolate is resistant to a drug or not. The sensitivity and specificity of the QFlu test will be calculated by comparing to the gold standard test.

ELIGIBILITY:
Inclusion Criteria:

* Those who exhibit flu-like symptom(s) during a flu season and who (or whose guardians) are willing to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There are three population of participants: pediatric (in patient or out patient), in-patient (any age) and out-patient (any age).
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2010-11-01; Primary Completion 2012-05-31 (Actual); Study Completion 2012-05-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for drug resistance detection | approximately 12 months after the study is completed.
  Interim results may be assessed after the first year study.

SECONDARY OUTCOMES:
Sensitivity and Specificity of the Test for Influenza Diagnosis | 12 months after the study is completed.
  Results may be assessed after the first year study.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland